CLINICAL TRIAL: NCT03058848
Title: A Study to Evaluate the Acceptability of a New Phenylalanine Free Infant Formula for Use in the Dietary Management of Phenylketonuria in Infants From Birth to 2 Year of Age With Regard to Product Tolerance and Adherence.
Brief Title: Evaluation of PKU Start
Acronym: PKU Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-PKUSTART-032016-29; 209920 (Registry Identifier: IRAS); 17/NW/0035 (Other: UK REC)
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonuria; Inborn Errors of Metabolism
Keywords: Phenylketonuria; PKU; Metabolism; Metabolic; Control; Acceptability
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumption of PKU Start (Experimental): Daily feed, substituting the participant's normal phe-free formula for PKU Start.
  Interventions: Dietary Supplement: PKU Start

INTERVENTIONS:
Dietary Supplement: PKU Start — PKU Start is a powdered, phenylalanine-free, infant formula, containing essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals, trace elements and long chain polyunsaturated fatty acids (LCPs); Arachidonic acid (AA) and Docosahexaenoic acid (DHA). It is suitable for use from birth.
  The recommended amount of the product for each participant will be determined and prescribed by a dietitian.

SUMMARY:
To evaluate the acceptability, tolerance and effect on metabolic control of PKU Start, a new Phe free protein substitute for the dietary management of PKU in infants from birth.

DETAILED DESCRIPTION:
This is an assessment of ten (10) infants who require a protein restricted diet that is low in Phe. Infants who routinely use a Phe free infant formula as part of their dietary therapy will be recruited for a 28-day assessment of PKU Start, to evaluate tolerance and acceptability.

The outcome of this assessment will be used in a submission to the regulatory authorities, Advisory Committee on Borderline Substances (ACBS), for PKU Start to become reimbursable on prescription in the UK.

The participant's dietitian will advise on an appropriate amount of PKU Start based on individual requirements. Parents/carers will be asked to substitute their usual Phe-free infant formula with PKU Start for one (1) month. The sponsor will supply PKU Start free of charge.

Prior to starting PKU Start, parents/carers will be asked to record information about the infant's usual GI tolerance and feeding pattern for a period of three (3) days, to allow for comparison between their existing formula and PKU Start.

They will be asked to record information about the following:

Stools Vomiting and Spit-up Feed / Fluid Intake and Compliance Phenylalanine Levels Final Evaluation about the presentation of the product, ease of preparation and how PKU Start flowed through the teat of a bottle.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of classical or severe PKU on new-born screening (For the purposes of this study, 'severe' is defined as phe concentrations between 120 and 600 µmol/L at diagnosis)
2. Taking a minimum of one (1) feed of a Phe-free infant formula
3. A minimum period of four (4) weeks from the time of diagnosis to initial approach to parents

Exclusion Criteria:

1. Diagnosed with mild PKU or hyperphenylalaninaemia (For the purposes of this study, 'mild' is defined as phe concentrations between 120 and 600 µmol/L at diagnosis)
2. Diagnosis of a congenital condition

Ages: 4 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Product compliance daily diary | Days 1-28
  Quantitative assessments from subject questionnaires that allow evaluation of compliance with the study product, i.e. actual versus prescribed intake.
GI tolerance daily diary | Days 1-28
  Qualitative assessments from subject questionnaires that allow evaluation of the gastro-intestinal tolerance of the study product.
Ease of use questionnaire | Day 29
  Qualitative assessment from subject questionnaire that allows evaluation of the ease of use of the study product.
Daily phenylalanine control | Days 1-28
  Collection of quantitative data regarding phenylalanine control using routine biochemical testing

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde, Glasgow, Lanarkshire
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided